CLINICAL TRIAL: NCT02036541
Title: A Prospective, Multicenter Clinical Trial Designed to Evaluate the Safety and Performance of the AqueSys XEN 45 Glaucoma Implant in Subjects With Refractory Glaucoma
Brief Title: AqueSys XEN 45 Glaucoma Implant in Refractory Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AqueSys, Inc. (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P13-001
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Glaucoma; Glaucoma, Open Angle
Keywords: Glaucoma Implant; Trabeculectomy; POAG; Primary Open Angle Glaucoma; Pseudoexfoliation Glaucoma; Pigmentary Glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Exfoliation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AqueSys XEN 45 Glaucoma Implant (Experimental)
  Interventions: Device: AqueSys XEN 45 Glaucoma Implant

INTERVENTIONS:
Device: AqueSys XEN 45 Glaucoma Implant — Placement of the AqueSys XEN 45 Glaucoma Implant in the study eye

SUMMARY:
To establish the safety and performance of the AqueSys XEN 45 Glaucoma Implant in eyes with refractory glaucoma.

DETAILED DESCRIPTION:
A prospective, multi-center, single arm, open-label clinical trial to evaluate the safety and IOP lowering performance of the AqueSys XEN 45 Glaucoma Implant in refractory glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Refractory Glaucoma
* Maximally-tolerated medicated IOP at two preoperative visits of ≥20 mmHg and ≤35 mmHg
* Visual field mean deviation score of -3 dB or worse
* Shaffer Angle Grade ≥ 3
* Area of free, healthy and mobile conjunctiva in the targeted quadrant

Exclusion Criteria:

* Active Neovascular Glaucoma
* Previous glaucoma shunt/valve in the targeted quadrant
* History of corneal surgery, opacities or disease/pathology
* Anticipated need for ocular surgery
* Non-study eye with BCVA of 20/200 or worse

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-01; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Lewis, M.D., Study Chair — Grutzmacher, Lewis & Sierra Surgical Eye Specialists
Locations (12):
- United States (12):
  - George R. Reiss, MD PC, Glendale, Arizona
  - Vold Vision, Fayetteville, Arkansas
  - Montebello Eye Center, Montebello, California
  - San Diego Eye Care Center, Oceanside, California
  - Palo Alto Eye Group, Palo Alto, California
  - Eye Center of Northern Colorado, Fort Collins, Colorado
  - Stiles Eyecare Excellence & Glaucoma Institute, Overland Park, Kansas
  - Washington University in St. Louis, Department of Ophthalmology, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Glaucoma Associates of Texas, Dallas, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - Spokane Eye Clinic, Spokane, Washington

REFERENCES:
- [Derived] Ozal SA, Kaplaner O, Basar BB, Guclu H, Ozal E. An innovation in glaucoma surgery: XEN45 gel stent implantation. Arq Bras Oftalmol. 2017 Nov-Dec;80(6):382-385. doi: 10.5935/0004-2749.20170093. PMID 29267575

RESULTS

PARTICIPANT FLOW:
Groups:
- XEN 45 Gel Stent: Placement of the XEN 45 Gel Stent in the study eye
Period: Overall Study
Arm/Group | XEN 45 Gel Stent
Started | 65
Completed Endpoint Visit | 54
Completed | 49
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | XEN 45 Gel Stent
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 65
Glaucoma Type [Count of Participants; unit: Participants]
  Primary Open Angle Glaucoma | 57
  Pseudoexfolative Glaucoma | 6
  Pigmentary Glaucoma | 1
  Mixed Mechanism Glaucoma | 1
Previous Cataract Surgery [Count of Participants; unit: Participants] | 45
Prior Glaucoma Procedure [Count of Participants; unit: Participants]
  Prior incisional glaucoma procedure | 41
  Prior laser trabeculoplasty | 14
  No prior glaucoma procedure | 10

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving a 20% or Greater Reduction in IOP From Baseline on the Same or Less Number of Medications
Description: Proportion of subjects achieving a 20% or greater reduction in IOP from baseline on the same or less number of medications. Subjects who underwent a glaucoma-related secondary surgical intervention prior to the 12-month visit were considered failures in this analysis.
Time Frame: 12 Months
Population: All subjects who completed the 12-month visit or underwent a glaucoma-related secondary surgical procedure prior to the 12-month visit were evaluated in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | XEN 45 Gel Stent
Number analyzed (Participants) | 61
Participants | 46

2. Primary Outcome: Mean Change in IOP From Baseline
Description: Mean change in IOP from baseline was calculated for subjects who completed the 12-month visit and the worst within-eye IOP was used for subjects who underwent a glaucoma-related secondary surgical intervention.
Time Frame: 12 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | XEN 45 Gel Stent
Number analyzed (Participants) | 61
mmHg | 6.2 (9.1)

ADVERSE EVENTS:
Time Frame: Ocular adverse events in the study are reported from the day of surgery (Day 0) through the 12-month visit
Description: Ocular adverse events in the study eye are reported from the day of surgery through the 12-month visit.
Arm/Group | XEN 45 Gel Stent
All-Cause Mortality (participants affected / at risk) | 2/65
Serious Adverse Events (participants affected / at risk) | 9/65
Other Adverse Events (participants affected / at risk) | 45/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XEN 45 Gel Stent (N=65)
Explant (Eye disorders) | 1 (1)
Secondary glaucoma procedure with explant (Eye disorders) | 6 (6)
Secondary glaucoma procedure (Eye disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XEN 45 Gel Stent (N=65)
Hypotony (IOP < 6 mmHg) (Eye disorders) | 16 (18) — All IOP < 6 mmHg was recorded as an adverse event, regardless of whether there were any associated complications or sequelae related to the low pressure. No clinically-significant consequences were associated with these hypotony cases
IOP increase ≥ 10 mmHg from baseline (Eye disorders) | 14 (18)
Needling procedure (Eye disorders) | 21 (29) — The protocol required these procedures to be recorded as adverse events
Wound dehiscence/leak (Eye disorders) | 6 (6)
Wound repair (Eye disorders) | 5 (6)
Anterior chamber tap (Eye disorders) | 6 (7)
Best-Corrected Visual Acuity Loss of ≥ 2 lines ≤ 30 days postop (Eye disorders) | 10 (10)
Best-Corrected Visual Acuity loss of ≥ 2 lines > 30 days (Eye disorders) | 7 (7)
Best-Corrected Visual Acuity loss of ≥ 2 lines at 12 Months (Eye disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the results of the multi-center trial must be published first, prior to any of the individual data being published